CLINICAL TRIAL: NCT03018496
Title: Investigating the Effects of Beta-Hydroxy-Beta-Methylbutyrate on Glucose Handling in Older and Younger Men.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: A12092016- ammendment 1
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2017-01

CONDITIONS: Insulin Resistance; Age Problems
MeSH Terms: conditions — Insulin Resistance | interventions — beta-hydroxyisovaleric acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Older Men (Experimental): Healthy male adults aged 18-35 Subjects will receive both HMB and placebo on separate visits in a crossover fashion
  Interventions: Dietary Supplement: Beta-Hydroxy-Beta-Methylbutyrate; Other: Placebo
- Younger Men (Experimental): Healthy male adults aged 65-85 Subjects will receive both HMB and placebo on separate visits in a crossover fashion
  Interventions: Dietary Supplement: Beta-Hydroxy-Beta-Methylbutyrate; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-Hydroxy-Beta-Methylbutyrate
  Other Names: HMB
Other: Placebo

SUMMARY:
This study intends to examine the effect of a commercially available nutritional supplement, Beta-hydroxy-beta-methylbutyrate(HMB) on whole-body responses to a sugar load.

DETAILED DESCRIPTION:
One change associated with human aging is a reduction in "fitness", both in terms of how far or quickly a person can run/cycle/swim and also in how well their blood vessels work. Additionally a person's metabolic fitness decreases; this is how well the body copes with nutrition and is why, for example, older people have a higher risk of diseases like type 2 diabetes. Previous studies have shown that as people become less fit, they are at increased risk of suffering a complication whilst undergoing surgery. It has also been shown that measuring how fit someone is, is better at predicting the risk of a surgical complication than purely using a person's age alone. Lots of research has shown that exercise can potentially reverse some of the age-related declines in fitness, however most has used long sessions of continuous exercise over a long period of time. High-intensity interval training (HIT), whereby people cycle on an exercise bike very hard for a minute, followed by a short rest, repeated over the course of 15 minutes can rapidly improve a person's fitness. However not everyone will be able to, or indeed want to participate in exercise this strenuous; therefore this research seeks to explore whether other options, such as dietary supplements can improve aspects of fitness

This study intends to examine the effect of giving a dietary supplement on the way a person's body handles the glucose (from carbohydrates/ sugars) in a meal. Previous work has shown that taking a beta-hydroxy beta-methyl butyrate (HMB) supplement may improve may improve a patient's response to glucose, however the evidence is not clear. HMB is a commercially available nutritional supplement providing a compound that the body produces each time protein is consumed, and is most commonly used by bodybuilders to help gain muscle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-35 or 65-85
* Male

Exclusion Criteria:

* Current participation in a formal exercise regime
* A BMI < 18 or > 32 kg·m2
* Active cardiovascular disease:

  o uncontrolled hypertension (BP > 160/100), angina, heart failure (class III/IV), Significant arrhythmia, right to left cardiac shunt, recent cardiac event
* Taking beta-adrenergic blocking agents,
* Cerebrovascular disease:

  o previous stroke, aneurysm (large vessel or intracranial), epilepsy
* Respiratory disease including:

  o pulmonary hypertension, significant COPD, uncontrolled asthma,
* Metabolic disease:

  o hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, type 1 or 2 diabetes
* Active inflammatory bowel or renal disease
* Malignancy
* Clotting dysfunction
* Significant musculoskeletal or neurological disorders
* Family history of early (<55y) death from cardiovascular disease

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Matsuda Index of insulin sensitivity | 180 minutes after a 75g oral glucose load
  Assessed from arterialised venous blood samples
Cederholm index of insulin sensitivity | 180 minutes after a 75g oral glucose load
  Assessed from arterialised venous blood samples

SECONDARY OUTCOMES:
Area-Under-Curve Glucose Concentration | 180 minutes after a 75g oral glucose load
  Assessed from arterialised venous blood samples
Area-Under-Curve Insulin Concentration | 180 minutes after a 75g oral glucose load
  Assessed from arterialised venous blood samples
Femoral Artery Blood flow | 15 minutes, 60 minutes and 120 minutes after a 75g oral glucose load
  Assessed using duplex ultrasonography of the superficial femoral artery of the right leg

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Nottingham, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510